CLINICAL TRIAL: NCT02675985
Title: Effects of Early Intensive Physical Therapy for Patients With Subarachnoid Hemorrhage in a Neurological ICU
Brief Title: Early Intensive Physical Therapy in Subarachnoid Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0829
Record Dates: First submitted 2016-02-02; First posted 2016-02-05 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Physical Therapy, early intervention
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Early intensive physical therapy will be the intervention arm. There is not a control group.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Early Intensive Physical therapy in the ICU

SUMMARY:
This study will investigate the safety and feasibility of early intensive physical therapy for patients diagnosed with subarachnoid hemorrhage. Intervention will begin in the neurological Intensive Care Unit (ICU) and continue for 30 days or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by CT scan or MRI with subarachnoid hemorrhage and admitted to the neurological ICU >48 hours.

Exclusion Criteria:

* Significant language barrier that would limit the ability to participate in the physical therapy program
* Severe baseline physical or cognitive impairment that would impair their ability to participate in the protocol
* Patients whose vital signs are outside the accepted starting and stopping criteria outlined below:

  1. intracranial pressure ≤ 15 mm Hg
  2. Cerebral perfusion pressure >50 or <70 mm Hg
  3. Mean arterial pressure ≥ 80 and ≤ 110
  4. Heart rate ≥40 and <140 bpm
  5. Pulse oximetry >88%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Improvement in Physical function in the ICU test (PFit) | Every 7 days until hospital discharge or 28 days of study enrollment

SECONDARY OUTCOMES:
Improvement in Activity Measure for Post-Acute Care (AM-PAC) mobility | Every 7 days until hospital discharge or 28 days of study enrollment
Improvement in Timed up and Go (TUG) | Every 7 days until hospital discharge or 28 days of study enrollment
Improvement in Postural Assessment Scale for Stroke Patients | Every 7 days until hospital discharge or 28 days of study enrollment
Improvement in Medical Research Council (MRC) Muscle Sum Score | Every 7 days until hospital discharge or 28 days of study enrollment
Improvement in Hand grip strength | Every 7 days until hospital discharge or 28 days of study enrollment

OTHER OUTCOMES:
Neuro-Quality of Life (QOL) | Hospital Discharge only
  Neuro-QOL measures 17 domains of health related quality of life for adults through self-report.. We will use the short form versions for applied cognition, lower extremity mobility and Upper extremity function and Satisfaction with social roles/activities.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Nordon-Craft, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCH, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moss M, Nordon-Craft A, Malone D, Van Pelt D, Frankel SK, Warner ML, Kriekels W, McNulty M, Fairclough DL, Schenkman M. A Randomized Trial of an Intensive Physical Therapy Program for Patients with Acute Respiratory Failure. Am J Respir Crit Care Med. 2016 May 15;193(10):1101-10. doi: 10.1164/rccm.201505-1039OC. PMID 26651376
- [Background] Sottile PD, Nordon-Craft A, Malone D, Schenkman M, Moss M. Patient and family perceptions of physical therapy in the medical intensive care unit. J Crit Care. 2015 Oct;30(5):891-5. doi: 10.1016/j.jcrc.2015.04.119. Epub 2015 May 8. PMID 26038155
- [Background] Denehy L, Nordon-Craft A, Edbrooke L, Malone D, Berney S, Schenkman M, Moss M. Outcome measures report different aspects of patient function three months following critical care. Intensive Care Med. 2014 Dec;40(12):1862-9. doi: 10.1007/s00134-014-3513-3. Epub 2014 Oct 16. PMID 25319384
- [Background] Nordon-Craft A, Schenkman M, Ridgeway K, Benson A, Moss M. Physical therapy management and patient outcomes following ICU-acquired weakness: a case series. J Neurol Phys Ther. 2011 Sep;35(3):133-40. doi: 10.1097/NPT.0b013e3182275905. PMID 21934375
- [Background] Olkowski BF, Devine MA, Slotnick LE, Veznedaroglu E, Liebman KM, Arcaro ML, Binning MJ. Safety and feasibility of an early mobilization program for patients with aneurysmal subarachnoid hemorrhage. Phys Ther. 2013 Feb;93(2):208-15. doi: 10.2522/ptj.20110334. Epub 2012 May 31. PMID 22652987